CLINICAL TRIAL: NCT04561193
Title: Investigation of Subsequent and Co-infections Associated With SARS-CoV-2 (COVID-19)
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 033.PHA.2020.A
Record Dates: First submitted 2020-09-22; First posted 2020-09-23 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective Cohort: Patients admitted to Methodist Richardson, Methodist Mansfield, Methodist Charlton, or Methodist Dallas Medical Centers between February 1, 2020 and April 30, 2020 with positive COVID-19 PCR test.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
Multicenter retrospective chart review of patients admitted to any of the four Methodist Health System hospitals

DETAILED DESCRIPTION:
Multicenter retrospective chart review of patients admitted to any of the four Methodist Health System hospitals (Methodist Richardson, Methodist Mansfield, Methodist Charlton, or Methodist Dallas) between February 1 and April 30, 2020. All study center utilize Epic ® electronic health record (Verona, Wisconsin; www.epic.com) for which all data will be extracted from.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Methodist Richardson, Methodist Mansfield, Methodist Charlton, or Methodist Dallas Medical Centers between February 1, 2020 and April 30, 2020
* >18 years old
* Positive SARS-CoV-2 (COVID-19) PCR test

Exclusion Criteria:

* Outpatient or emergency department visit
* Not admitted to an inpatient or observation status for >24 hours

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with positive COVID-19 PCR test admitted to Methodist Richardson, Methodist Mansfield, Methodist Charlton, or Methodist Dallas Medical Centers between February 1, 2020 and April 30, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Prevalence of subsequent and co-infections | Feb 2020 - April 2020
  Prevalence of subsequent and co-infections

SECONDARY OUTCOMES:
In-hospital mortality | Feb 2020 - April 2020
  In-hospital mortality
Hospital length of stay (LOS) | Feb 2020 - April 2020
  Hospital length of stay (LOS)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Crotty, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No